CLINICAL TRIAL: NCT06272799
Title: Tolerability and Efficacy of Adjuvant T-DM1 in Patients with HER2 Positive Breast Cancer After Incomplete Pathological Response to Neoadjuvant Chemotherapy Including Anti-HER2 Agents. Real-world Multicenter Retrospective-prospective Study. ATD-Study.
Brief Title: Tolerability and Efficacy of Adjuvant T-DM1 in Patients with HER2 Positive Breast Cancer After Incomplete Pathological Response to Neoadjuvant Chemotherapy Including Anti-HER2 Agents.
Acronym: ATD
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS1480/21
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective cohort: 80 patients will form the retrospective cohort, considering consecutively all patients treated according to clinical practice outside of studies randomized
  Interventions: Drug: T-DM1 adjuvant
- Prospectively cohort: Additional 80 patients who meet the inclusion criteria will be enrolled prospectively
  Interventions: Drug: T-DM1 adjuvant

INTERVENTIONS:
Drug: T-DM1 adjuvant — Evaluate the tolerability of treatment with adjuvant T-DM1 after failure to respond complete pathology to neoadjuvant treatment in terms of adverse events

SUMMARY:
Multicenter, retrospective-prospective, real-world observational study, with the aim of evaluating tolerability and efficacy in a population of patients treated according to clinical practice outside of studies randomized.

DETAILED DESCRIPTION:
Patients affected by will be included in the study and analyzed HER2 positive breast cancer with residual invasive disease after neoadjuvant chemotherapy, treated consecutively with adjuvant T-DM1 at the various Italian oncology centers.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of HER2 positive breast cancer;
* Presence of invasive residual disease on T or N after neoadjuvant chemotherapy including anti-HER2 agents
* Treatment with T-DM1 in the adjuvant post-neoadjuvant setting, in case of positive hormone receptors in combination with adjuvant hormone therapy. Complementary radiotherapy will be allowed as per lines guide;
* Availability of adequate information regarding treatment with adjuvant T-DM1 in accordance with the objectives of the study;
* Written informed consent for the prospective part and, if possible, for the recruited patients retrospectively

Exclusion Criteria:

* Concomitant treatments with other biological agents;
* Absence of clinical data that allow the correct analysis of the primary and secondary objectives;
* Patients with a history of other malignant neoplasms;
* Contraindications to the use of T-DM

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HER2 positive breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Evaluate the tolerability. | 24 months
  Evaluate the tolerability of the treatment in terms of adverse events, defined according to Common Terminology Criteria for Adverse Events (CTCAE, version 4), in a population of patients treated with adjuvant T-DM1 in "real life"

SECONDARY OUTCOMES:
Evaluate the effectiveness of treatment. | 24 months
  Evaluate in the "real life setting" the effectiveness of adjuvant treatment in terms of survival free from disease (Disease Free Survival, DFS) in patients with HER2 positive breast cancer and residual invasive disease (on T and/or on N) after neoadjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No